CLINICAL TRIAL: NCT02119364
Title: Computer Based Working Memory Training in Children With Cerebral Palsy (CP)
Brief Title: Working Memory Training for Children With Cerebral Palsy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sorlandet Hospital HF (Other Government)
Collaborators: Helse Sor-Ost (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2012/2/00|14
Record Dates: First submitted 2013-04-03; First posted 2014-04-21 (Estimated); Last update posted 2014-04-21 (Estimated); Status verified 2014-04

CONDITIONS: Cerebral Palsy
Keywords: cerebral palsy; working memory; cognitive training
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Working memory training (Active Comparator): After baseline assessment participants will be randomized to active training or treatment as usual (waiting). The active group will start training immediately and will have 6 weeks to perform the 25 training sessions.
  Interventions: Other: Working memory training
- Passive control group (No Intervention): The control group will receive "treatment as usual" (special education, physiotherapy etc).

INTERVENTIONS:
Other: Working memory training — The child will use the computer program at home under parental supervision for 25 sessions, each lasting 30-45 minutes and the family has 6 weeks to complete the training. Each session consists of 8 different tasks presented by an animated robot. The tasks all require the child to hold information in working memory and to manipulate the information.
  Other Names: Cogmed RoboMemo
  Arms: Working memory training

SUMMARY:
Cerebral palsy (CP) is the most common motor disability in childhood (2-3 per 1000 live born), and is frequently accompanied by cognitive impairments and behavioural problems. The present study is a controlled clinical trial, a multicenter-study involving three health regions, as well as the Norwegian University of Science and Technology (NTNU). Its primary research goal will be to evaluate the effects of computer-based cognitive training in children with CP. In addition, this study will be the first to conduct a comprehensive neuropsychological examination to improve our understanding of cognitive impairments as well as cognitive resources in CP children in Norway to aid in intervention planning.

ELIGIBILITY:
Inclusion Criteria:

* Cerebral Palsy
* School age (7-15 years of age)

Exclusion Criteria:

* Not able to use computer, blind, deaf

Ages: 7 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 115 (Estimated)
Dates: Start 2013-10; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Spatial span | 9-12 weeks after inclusion
  The spatial span board from the Wechsler Memory scale 3ed. will represent our primary outcome measure. The total of forward and backward span will be used as primary outcome measure.

SECONDARY OUTCOMES:
Verbal working memory | 9-12 weeks after inclusion
  The sum of letter-number sequencing and digit span (total raw scores) will be used as secondary outcome measures.

OTHER OUTCOMES:
Attention Deficit Hyperactivity Disorder rating scale | 9-12 weeks after inclusion
  To assess changes in symptoms of attention/hyperactivity problems after training.
Activity of daily life | 9-12 weeks after inclusion
  Vineland adaptive behaviour scale is a semi-structured parental interview assessing daily life functioning.
Attention/executive functions assessed by parents | 9-12 weeks after inclusion
  BRIEF is a parental questionnaire that assesses aspects of attention and executive function in daily life.

CONTACTS AND LOCATIONS:
Overall Officials: Gro CC Lohaugen, Phd, Principal Investigator — Department of Child rehabilitation, Sørlandet Hospital, Arendal, Norway
Locations (1):
- Sorlandet Hospital, Arendal, Aust-Agder, Norway

REFERENCES:
- [Derived] Lohaugen GC, Beneventi H, Andersen GL, Sundberg C, Ostgard HF, Bakkan E, Walther G, Vik T, Skranes J. Do children with cerebral palsy benefit from computerized working memory training? Study protocol for a randomized controlled trial. Trials. 2014 Jul 7;15:269. doi: 10.1186/1745-6215-15-269. PMID 24998242